CLINICAL TRIAL: NCT00814658
Title: The Use of Galantamine (Reminyl ER) in Patients With MIXed Dementia: Effects on Cognition and Quality of Life
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag Farmaceutica Ltda. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR014938; GALDEM4008 (Other: Janssen-Cilag Farmaceutica Ltda.)
Record Dates: First submitted 2008-12-24; First posted 2008-12-25 (Estimated); Results first posted 2013-08-26 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Dementia
Keywords: Dementia; Mixed Dementia; Galantamine; Reminyl ER; Nimodipine
MeSH Terms: conditions — Dementia; Mixed Dementias | interventions — Galantamine; Nimodipine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Galantamine + Nimodipine (Experimental)
  Interventions: Drug: Galantamine; Drug: Nimodipine
- Galantamine + Placebo (Experimental)
  Interventions: Drug: Galantamine; Drug: Placebo

INTERVENTIONS:
Drug: Galantamine — Galantamine 8 mg/day for one month, followed by 4 weeks of galantamine 16 mg/day. If necessary and well tolerated, dosage of galantamine will be increased to 24 mg/day.
Drug: Nimodipine — Nimodipine 30 mg 3 times a day (tid).
  Arms: Galantamine + Nimodipine
Drug: Placebo — Matching placebo three times a day (tid).
  Arms: Galantamine + Placebo

SUMMARY:
The purpose of this study is to evaluate the combination of galantamine with nimodipine in patients with mixed dementia on cognition and quality of life.

DETAILED DESCRIPTION:
A double-blind (neither the patient nor the physician know the name of the study drug), 6-month, multicenter, placebo-controlled trial to evaluate the combination of galantamine with nimodipine in patients with mixed dementia on cognition and quality of life. The target dose of galantamine is 24 mg/day and nimodipine will be taken in fixed doses of 90 mg/day. Primary outcomes will be measured by a computerized battery of neuropsychological tests and Quality of Life (QoL) scores. Secondary outcomes will be measured by ADAS-cog, Clinical Global Impression (CGI) and Neuropsychiatric Inventory (NPI). Mixed dementia (Alzheimer's Disease (AD) associated with cerebrovascular disease) is one of the most common causes of dementia, which remain largely underdiagnosed. Little is known about specific treatments for this condition. Ischemic lesions by themselves seem to play an important role in cognitive impairment, even in the presence of AD pathology. Hypotheses: - Galantamine 16-24 mg/day in combination with nimodipine 90 mg/day is superior to galantamine monotherapy (16-24 mg/day) in improving or stabilizing cognition in patients with AD associated with cerebrovascular disease (mixed dementia), as measured by the CNTB at 6 months. - Galantamine 16-24 mg/day in combination with nimodipine 90 mg/day is superior to galantamine monotherapy (16-24 mg/day) on QoL measures in this population as measured by QoL - AD at 6 months. Group 1: galantamine oral 8mg/day for a month, 16mg/day for 4 weeks and after 24mg/day until end of study plus nimodipine oral 30mg tid during all study. Group 2: Group 1: galantamine oral 8mg/day for a month, 16mg/day for 4 weeks and after 24mg/day until end of study plus placebo oral 30mg tid during all study.

ELIGIBILITY:
Inclusion Criteria:

* Patients should fulfill DSM-IV criteria for dementia (APA, 1994)
* Patients should fulfill criteria for AD with cerebrovascular disease according to NINDS-AIREN criteria (Román et al., 1993)
* The severity of dementia should be mild to moderate, as defined by MMSE score between 10 and 26 (inclusive)
* Patients (and their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

* History of neurodegenerative disorders such as Parkinson's disease, Pick's disease or Huntington's chorea, Down's syndrome, Creutzfeldt-Jacob disease. Patients who have mild extrapyramidal signs, for which no treatment is required, are not excluded from the trial
* History of liver or renal insufficiency
* significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurological, psychiatric, or metabolic disturbances in the past 6 months
* Patients who have previously received M1 agonists or cholinesterase inhibitors (tacrine, donepezil, metrifonate, rivastigmine) for treatment of Alzheimer's disease, no matter if approved or experimental can be included in this trial provided there was at least a washout period of 60 days prior to the screening assessments
* History of drug or alcohol abuse within the last year or prior prolonged history
* History of severe drug allergy or hypersensitivity
* including recorded hypersensitivity to cholinesterase inhibitors, choline agonists or similar agents, or bromide
* Subjects who have previously been enrolled in other galantamine trials.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Farmaceutica Ltda. Clinical Trial, Study Director — Janssen-Cilag Farmaceutica Ltda.

REFERENCES:
- [Derived] Caramelli P, Laks J, Palmini AL, Nitrini R, Chaves ML, Forlenza OV, Vale Fde A, Barbosa MT, Bottino CM, Machado JC, Charchat-Fichman H, Lawson FL. Effects of galantamine and galantamine combined with nimodipine on cognitive speed and quality of life in mixed dementia: a 24-week, randomized, placebo-controlled exploratory trial (the REMIX study). Arq Neuropsiquiatr. 2014 Jun;72(6):411-7. doi: 10.1590/0004-282x20140055. PMID 24964105

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 22 patients were enrolled in the study, but one (1) patient was excluded from the study because the patient has died before study medication use. Therefore, the study was formed by 21 patients that used at least 1 study medication dose and had at least 1 evaluation after started use (Intention to Treat (ITT) population).
Groups:
- Galantamine + Nimodipine: Galantamine 8 mg/day for one month + nimodipine 30 mg 3 times a day (tid), followed by 4 weeks of galantamine 16 mg/day + nimodipine 30 mg tid. If necessary and well tolerated, dosage of galantamine will be increased to 24 mg/day + nimodipine 30 mg tid.
- Galantamine + Placebo: Galantamine 8 mg/day and placebo three times a day (tid) for 4 weeks, followed by 4 weeks of galantamine 16 mg/day and placebo tid. If necessary and well tolerated, galantamine dosage may be increased to 24 mg/day, together with placebo tid.
Period: Overall Study
Arm/Group | Galantamine + Nimodipine | Galantamine + Placebo
Started | 9 | 12
Completed | 5 | 8
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Galantamine + Nimodipine | Galantamine + Placebo | Total
Number analyzed (Participants) | 9 | 12 | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 78.1 (5.3) | 74.3 (6.5) | 76.0 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Reaction Time for Simple Reaction Time Test at Baseline, Week 8, and Week 24
Description: The Simple Reaction Time is a computerized attention test that evaluates the patient's reaction time. The number one was presented in the center of the computer screen and the patient had to press this number in the response box as quickly as possible. The reaction time, assessed 100 times per patient, was averaged at each time point for each patient e.g., at baseline, Week 8 and Week 24. The patient's finger was put over button one before the test begun. This test is part of the Computerized Neuropsychological Test Battery (CNTB).
Time Frame: Baseline, Week 8, Week 24
Population: Intent to Treat population, which consisted of all participants who used at least 1 study medication dose, had at least 1 evaluation after started use, and with evaluable data at each measurement time point.
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Galantamine + Nimodipine (Baseline); Galantamine + Nimodipine (Week 8); Galantamine + Nimodipine (Week 24): Galantamine 8 mg/day for one month + nimodipine 30 mg 3 times a day (tid), followed by 4 weeks of galantamine 16 mg/day + nimodipine 30 mg tid. If necessary and well tolerated, dosage of galantamine will be increased to 24 mg/day + nimodipine 30 mg tid.
- Galantamine + Placebo (Baseline); Galantamine + Placebo (Week 8); Galantamine + Placebo (Week 24): Galantamine 8 mg/day and placebo three times a day (tid) for 4 weeks, followed by 4 weeks of galantamine 16 mg/day and placebo tid. If necessary and well tolerated, galantamine dosage may be increased to 24 mg/day, together with placebo tid.
Arm/Group | Galantamine + Nimodipine (Baseline) | Galantamine + Placebo (Baseline) | Galantamine + Nimodipine (Week 8) | Galantamine + Placebo (Week 8) | Galantamine + Nimodipine (Week 24) | Galantamine + Placebo (Week 24)
Number analyzed (Participants) | 9 | 12 | 5 | 9 | 5 | 8
milliseconds | 1024.06 (1307.97) | 729.18 (394.88) | 466.60 (297.53) | 671.33 (298.38) | 467.60 (336.69) | 584.44 (320.37)

2. Primary Outcome: Reaction Time for Two-choice Reaction Time Test at Baseline, Week 8, and Week 24
Description: The Two-choice reaction time test is a computerized attention test in which the numbers one or five were presented in the center of the computer screen in a random order. The patient had to press the correspondent button in the response box as quickly as possible. The patient's right finger was put over the button five and the left finger over button one before the test begun. The reaction time, assessed 100 times per patient, was averaged at each time point for each patient e.g., at baseline, Week 8 and Week 24.This test is part of the Computerized Neuropsychological Test Battery (CNTB).
Time Frame: Baseline, Week 8, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Galantamine + Nimodipine (Baseline) | Galantamine + Placebo (Baseline) | Galantamine + Nimodipine (Week 8) | Galantamine + Placebo (Week 8) | Galantamine + Nimodipine (Week 24) | Galantamine + Placebo (Week 24)
Number analyzed (Participants) | 9 | 12 | 5 | 9 | 5 | 8
milliseconds | 1919.72 (1801.13) | 1096.75 (617.45) | 852.70 (480.79) | 1187.78 (637.60) | 727.60 (375.03) | 1116.25 (540.91)

3. Primary Outcome: Reaction Time for Face Recognition Test at Baseline, Week 8, and Week 24
Description: The face recognition test is a computerized attention test in which ten unfamiliar faces were presented simultaneously on the computer screen for ten seconds to be remembered. After that, a single face was shown and the patient had to press the button one if he/she remembered or, otherwise, button five. It consisted of a random presentation of ten pre-exposed faces and ten new faces as distracters. The reaction time, assessed per patient, was averaged at each time point for each patient e.g., at baseline, Weeks 8 and 24. This test is part of the Computerized Neuropsychological Test Battery.
Time Frame: Baseline, Week 8, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Galantamine + Nimodipine (Baseline) | Galantamine + Placebo (Baseline) | Galantamine + Nimodipine (Week 8) | Galantamine + Placebo (Week 8) | Galantamine + Nimodipine (Week 24) | Galantamine + Placebo (Week 24)
Number analyzed (Participants) | 9 | 12 | 5 | 9 | 5 | 8
milliseconds | 3124.00 (1461.46) | 2684.45 (1315.44) | 2262.50 (803.30) | 2734.25 (1252.62) | 2357.80 (1919.72) | 3099.38 (1823.80)

4. Primary Outcome: Reaction Time for Word Recognition and Learning Test at Baseline, Week 8, and Week 24
Description: The reaction time for word recognition and learning test is a computerized attention test that evaluates the patient's reaction time. This test is similar to the Face Recognition test procedure using Words. The recognition procedure was repeated three times to evaluate a learning effect. The reaction time, assessed per patient, was averaged at each time point for each patient e.g., at baseline, Week 8 and Week 24. This test is part of the Computerized Neuropsychological Test Battery (CNTB).
Time Frame: Baseline, Week 8, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Galantamine + Nimodipine (Baseline) | Galantamine + Placebo (Baseline) | Galantamine + Nimodipine (Week 8) | Galantamine + Placebo (Week 8) | Galantamine + Nimodipine (Week 24) | Galantamine + Placebo (Week 24)
Number analyzed (Participants) | 9 | 12 | 5 | 9 | 5 | 8
milliseconds | 2022.17 (672.08) | 2978.77 (1867.62) | 1966.40 (1252.10) | 2379.83 (984.52) | 1722.00 (1174.22) | 3038.81 (1243.79)

5. Primary Outcome: The Quality of Life Assessment for Caregivers of Patients With Alzheimer's Disease (QoL- AD) Total Scores at Baseline, Week 8, Week 24
Description: The Quality of Life assessment scale for caregivers of patients with Alzheimer's disease (QoL-AD) is a 13-item scale with four possible scores for each question (score 1: poor and score 4: excellent). It evaluates the caregivers own perceived quality of life. Total score ranges from 13 to 52. Higher scores represent a better outcome.
Time Frame: Baseline, Week 8, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Galantamine + Nimodipine (Baseline) | Galantamine + Placebo (Baseline) | Galantamine + Nimodipine (Week 8) | Galantamine + Placebo (Week 8) | Galantamine + Nimodipine (Week 24) | Galantamine + Placebo (Week 24)
Number analyzed (Participants) | 9 | 12 | 5 | 9 | 5 | 8
scores on a scale | 34.00 (6.98) | 36.50 (7.40) | 32.00 (9.03) | 33.56 (6.84) | 36.60 (4.56) | 34.88 (6.83)

6. Primary Outcome: The Quality of Life Assessment for Patients With Alzheimer's Disease (QoL- AD) Total Scores at Baseline, Week 8, Week 24
Description: The Quality of Life assessment scale for patients with Alzheimer's disease (QoL-AD) is a 13-item scale with four possible scores for each question (score 1: poor and score 4: excellent). Total score ranges from 13 to 52. Higher scores represent a better outcome.
Time Frame: Baseline, Week 8, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Galantamine + Nimodipine (Baseline) | Galantamine + Placebo (Baseline) | Galantamine + Nimodipine (Week 8) | Galantamine + Placebo (Week 8) | Galantamine + Nimodipine (Week 24) | Galantamine + Placebo (Week 24)
Number analyzed (Participants) | 9 | 12 | 5 | 9 | 5 | 7
scores on a scale | 33.56 (5.59) | 32.67 (7.02) | 35.60 (3.71) | 33.11 (4.68) | 36.60 (6.23) | 33.86 (5.27)

7. Primary Outcome: The Quality of Life Assessment for Patients With Alzheimer's Disease (QoL- AD) Total Scores, Based on the Caregiver's Opinion, at Baseline, Week 8, Week 24
Description: The Quality of Life assessment scale for patients with Alzheimer's disease (QoL-AD), according to the opinion of the caregiver is a 13-item scale with four possible scores for each question (score 1: poor and score 4: excellent). It evaluates the opinion of the caregiver about the patient's quality of life. Total score ranges from 13 to 52. Higher scores represent a better outcome.
Time Frame: Baseline, Week 8, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Galantamine + Nimodipine (Baseline) | Galantamine + Placebo (Baseline) | Galantamine + Nimodipine (Week 8) | Galantamine + Placebo (Week 8) | Galantamine + Nimodipine (Week 24) | Galantamine + Placebo (Week 24)
Number analyzed (Participants) | 9 | 12 | 5 | 9 | 5 | 8
scores on a scale | 28.33 (8.62) | 29.33 (8.08) | 27.80 (5.36) | 29.78 (6.69) | 29.80 (5.76) | 29.13 (7.00)

8. Secondary Outcome: The Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog) at Baseline, Week 8, and Week 24
Description: The ADAS-Cog is a psychometric instrument that evaluates memory, attention, reasoning, language, orientation and praxis using an 11-point Assessment Scale. It has a minimum score of 0 and a maximum severity score of 70, and a higher score indicates more impairment.
Time Frame: Baseline, Week 8, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Galantamine + Nimodipine (Baseline) | Galantamine + Placebo (Baseline) | Galantamine + Nimodipine (Week 8) | Galantamine + Placebo (Week 8) | Galantamine + Nimodipine (Week 24) | Galantamine + Placebo (Week 24)
Number analyzed (Participants) | 9 | 11 | 5 | 9 | 5 | 8
scores on a scale | 30.40 (13.81) | 28.20 (11.06) | 25.10 (9.21) | 31.03 (11.45) | 25.02 (9.75) | 27.70 (12.16)

9. Secondary Outcome: The Clinical Global Impression (CGI) at Week 4, Week 8, Week 16, and Week 24
Description: The Clinical Global Impression (CGI) is a scale to assess treatment response in patients with mental disorders. The Clinical Global Impression Improvement scale (CGI-I) requires the clinician to rate how much the patient's illness has improved or worsened relative to a baseline state. A patient's illness is compared to change over time and rated as: very much improved, much improved, minimally improved, no change, minimally worse, much worse, or very much worse.
Time Frame: Week 4, Week 8, Week 16, Week 24
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Galantamine + Nimodipine (Week 4); Galantamine + Nimodipine (Week 8); Galantamine + Nimodipine (Week 16); Galantamine + Nimodipine (Week 24): Galantamine 8 mg/day for one month + nimodipine 30 mg 3 times a day (tid), followed by 4 weeks of galantamine 16 mg/day + nimodipine 30 mg tid. If necessary and well tolerated, dosage of galantamine will be increased to 24 mg/day + nimodipine 30 mg tid.
- Galantamine + Placebo (Week 4); Galantamine + Placebo (Week 8); Galantamine + Placebo (Week 16); Galantamine + Placebo (Week 24): Galantamine 8 mg/day and placebo three times a day (tid) for 4 weeks, followed by 4 weeks of galantamine 16 mg/day and placebo tid. If necessary and well tolerated, galantamine dosage may be increased to 24 mg/day, together with placebo tid.
Arm/Group | Galantamine + Nimodipine (Week 4) | Galantamine + Placebo (Week 4) | Galantamine + Nimodipine (Week 8) | Galantamine + Placebo (Week 8) | Galantamine + Nimodipine (Week 16) | Galantamine + Placebo (Week 16) | Galantamine + Nimodipine (Week 24) | Galantamine + Placebo (Week 24)
Number analyzed (Participants) | 7 | 10 | 5 | 9 | 5 | 8 | 5 | 8
participants
  Very much improved | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Much improved | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 2
  Minimally improved | 1 | 5 | 2 | 6 | 2 | 3 | 3 | 4
  No change | 4 | 4 | 2 | 2 | 1 | 5 | 1 | 1
  Minimally worse | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
  Much worse | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Very much worse | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: The Neuropsychiatric Inventory (NPI) at Baseline, Week 8, and Week 24
Description: The NPI evaluates 12 neuropsychiatric domains: delusions, hallucinations, dysphoria, anxiety, aggression, euphoria, dis-inhibition, irritability/lability, apathy, aberrant motor activity, eating disorders, and night-time behavior disturbances. For present domains, the severity and frequency of the behavior are determined. Frequency is rated 1 (rarely) to 4 (very often) and Severity is scored 1 (mild) to 3 (severe). The product scores vary from 1 (mild and rarely) to 12 (very often and severe). Total scores vary from 0 (no present domain) to 144 (all domains are present, are often and severe).
Time Frame: Baseline, Week 8, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Galantamine + Nimodipine (Baseline) | Galantamine + Placebo (Baseline) | Galantamine + Nimodipine (Week 8) | Galantamine + Placebo (Week 8) | Galantamine + Nimodipine (Week 24) | Galantamine + Placebo (Week 24)
Number analyzed (Participants) | 9 | 12 | 5 | 12 | 5 | 8
scores on a scale | 24.0 (14.72) | 26.92 (20.66) | 20.20 (8.67) | 22.11 (17.93) | 15.00 (11.55) | 19.75 (16.58)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Galantamine + Nimodipine | Galantamine + Placebo
Serious Adverse Events (participants affected / at risk) | 1/9 | 1/12
Other Adverse Events (participants affected / at risk) | 8/9 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Galantamine + Nimodipine (N=9) | Galantamine + Placebo (N=12)
Fall (Injury, poisoning and procedural complications) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Galantamine + Nimodipine (N=9) | Galantamine + Placebo (N=12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Tinnitus (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 2
Sleepiness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2
Vertigo (Nervous system disorders) | 0 | 1
Gastrointestinal anomaly (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Dry lips (Gastrointestinal disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 2 | 3
Blood glucose floating (Investigations) | 1 | 0
Loss weight (Investigations) | 1 | 0
Murmur (Investigations) | 1 | 0
Respiratory airways bacterial infection (Infections and infestations) | 1 | 0
Upper respiratory airways viral infection (Infections and infestations) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 1
Aggressiveness (Psychiatric disorders) | 3 | 0
Visual hallucination (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Impatience (Psychiatric disorders) | 0 | 1
Irritability (Psychiatric disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Flu symptoms (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 1
Nervousness (General disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The major limitation of this study was the small sample size. This was probably due to the short enrollment period and to the rigorous inclusion criteria that were adopted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor can require changes to the communication and can extend the embargo.